CLINICAL TRIAL: NCT07110896
Title: A Randomized, Placebo-controlled, Double-blind Clinical Study to Evaluate the Effect of Humiome® Post LB on Stress, Anxiety, and Cognition in Aging Adults
Brief Title: Study Evaluating the Effect of Humiome® Post LB on Stress, Anxiety, and Cognition in Aging Adults
Acronym: AnexLB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: Analyze & Realize (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2024-09-06-ANEX
Record Dates: First submitted 2025-06-19; First posted 2025-08-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-06

CONDITIONS: Healthy Aging
Keywords: Healthy aging; Microbiome; Stress; Sleep; Anxiety; gut-brain
MeSH Terms: conditions — Anxiety Disorders | interventions — Lacteol; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Parallel Assignment A randomized, placebo-controlled, double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Humiome Post LB (Postbiotic) : 340mg in 2 identical capsules per day orally
  Interventions: Dietary Supplement: Humiome Post LB (Postbiotic)
- Placebo (Placebo Comparator): Microcrystalline in 2 identical capsules per day orally
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Humiome Post LB (Postbiotic) — Heat-inactivated lactobacilli with fermented medium (a postbiotic) in 340mg powder format
  Other Names: Lactobacillus LB
  Arms: Active
Dietary Supplement: Placebo — Microcrystalline cellulose, 340mg powder format
  Other Names: microcrystalline cellulose
  Arms: Placebo

SUMMARY:
To assess the effect of 3 months of daily consumption of a postbiotic (inactivated lactic acid bacteria) Humiome® Post LB on stress measured by the Depression Anxiety Stress Scale-21 (DASS-21) adjusted on baseline in study participants when compared to placebo

DETAILED DESCRIPTION:
A double-blinded, randomised and placebo-controlled study will be conducted to assess the effect of 3 months of daily consumption of a postbiotic (inactivated lactic acid bacteria), Humiome® Post LB, on stress measured by the Depression Anxiety Stress Scale-21 (DASS-21) adjusted for baseline in study participants when compared to placebo.

The study will be in healthy subjects who are getting older (ageing population) and will measure factors such as stress, sleep, anxiety as well as gut microbiome. The intervention period will be 90 days, and study will include 236 subjects in two arms (active and placebo),

ELIGIBILITY:
Inclusion Criteria

1. Participant is male or female, 50-75 years of age, inclusive.
2. Participant has a Body Mass Index (BMI) of ≥18.5 kg/m2 to 32 kg/m2.
3. Participant is generally in good health, as per investigator's judgement at V1.
4. Participant has subjective mild to moderate memory complaints, as per investigator's judgement.
5. Participant has a total score of ≥42 and ≤60 on the DASS-21 administered at V1.
6. Participant is willing to maintain regular dietary, exercise, and allowed medication/supplement habits and smoking and other nicotine habits (if a smoker or nicotine user) for the duration of the study.
7. Participant understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study investigator.

7. Participant understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study investigator.

Exclusion criteria:

1. Participant has a history or presence of a psychiatric or neurologic disease including epilepsy, cerebrovascular disease, traumatic brain injury, dementia, Alzheimer's Disease, clinical depression, or other clinically significant psychiatric/neurologic condition that, in the opinion of the investigator, could interfere with the interpretation of the study results.
2. MMSE score at V1 < 21.
3. Chronic fatigue syndrome.
4. Women: elevated stress and/or anxiety levels clearly related to the (peri) menopause complaints, as per investigator judgement
5. Non-pharmacological or non-supplementation options for management of stress, anxiety or memory/cognitive complaints (e.g. yoga, "brain jogging") started within 4 weeks of screening 6. Participant has a clinically significant gastrointestinal, endocrine, cardiovascular, renal, hepatic, pulmonary, pancreatic, neurologic, or biliary disorder that, in the opinion of the investigator, could interfere with the interpretation of the study results.

7. Participant has a condition that would likely cause immunosuppression. 8. Participant has a history of gastrointestinal surgery (cholecystectomy and appendectomy are acceptable, considering the prevalence in the age group), as per investigator judgement. 9. Participant has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg) at screening.

10. Participant has an issue with hearing or seeing that might interfere with the tasks/questionnaires to be completed during the visits.

11. Participant has used pre-, pro-, syn-, or post-biotic supplements within 90 days of screening.

12. Participant has a history of using psychotropic medications (including antidepressants and tranquilizers), stimulant medications, and/or narcotics within 4 weeks of screening. 13. Participants has major sleep disorder (severe insomnia) based on investigator's judgment.

14. Participant has used sleep aid medications, supplements, and/or products, including antihistamines, within 2 weeks of screening (washout prior to screening is allowed). Sporadic use of supplementation of melatonin, valerian, passion flower, lavender, if needed, if this has been habitually or occasionally done prior to the study, is allowed. 15. Participant has used an acid-blocking medication (e.g., proton pump inhibitor, H2 blocker) in the past 30 days prior to study. However, any ongoing use started at least 12 weeks before Visit 1 is allowed.

16. Participant has used selective serotonin reuptake inhibitors (SSRIs) or benzodiazepines in the past 30 days. (Note: Participants will not be excluded on the basis of a well-managed depressive disorder that does not require SSRIs.) 17. Participant has a history of cancer in the prior 5 years. 18. Participant has an allergy to any components of the IP or the standardized breakfast.

19. Individual has signs or symptoms of an active infection of clinical significance or has taken antibiotics within 30 days prior to any visit (washout is permitted for re-scheduling of the clinic visit).

20. Participant has been exposed to any non-registered drug product within 30 days of the screening visit.

21. Participant has a current or recent history (within 12 months of screening) or strong potential for illicit drug or excessive alcohol intake defined as >14 drinks per week (1 drink = 350 ml beer, 150 ml wine, or 40 ml hard liquor).

22. Women lactating, pregnant or of childbearing potential not using a reliable contraceptive method.

23. Participant has a condition the investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Effect on stress | Timeframe - Day 0 (V2), and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on stress measured by the Depression Anxiety Stress Scale-21 (DASS-21) adjusted on baseline in study participants when compared to placebo

SECONDARY OUTCOMES:
Effect on stress (adjusted to baseline) | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on stress measured by the Depression Anxiety Stress Scale-21 (DASS-21) adjusted on baseline in study participants when compared to placebo. Lowest Value: 0, Highest Value: 42. A higher score means a worse outcome
Effect on stress (within the group) | (Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on change in DASS-21 subscores of stress, depression, anxiety in study participants when compared to placebo (between group comparison) and baseline (withingroup comparison). Lowest Value: 0, Highest Value: 42. A higher score means a worse outcome
Effect on stress (within the group, compared to baseline) | (Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB and Placebo on stress measured by the DASS-21 in study participants when compared to baseline. Lowest Value: 0, Highest Value: 42. A higher score means a worse outcome.
Effect on indicators of Anxiety | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on indicators of anxiety when compared to placebo and baseline . The GAD-7 total score (range 0-21, expressed in a.u.) will be used to assess indicators of anxiety. Lowest Value: 0 Highest Value: 21. A higher score means a worse outcome
Effect on indicators of perceived stress | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on indicators of perceived stress when compared to placebo and baseline. The PSS-10 total score (range 0-40; expressed in a.u.) will be used to assess indicators of perceived stress. Lowest Value: 0, Highest Value: 40. A higher score means a worse outcome,
Effect on Indicators of cognition and memory | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on indicators of Indicators of cognition and memory when compared to placebo and baseline. Cogstate International Digit Symbol Substitution Test (symbols) will be used to test domains processing speed test, assesses focused attention and aspects of executive functioning; the outcome is the total number of correct responses
Effect on indicators of Chronic inflammation (hs-CRP) in blood | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on indicators of Chronic inflammation in blood when compared to placebo and baseline. For this hs-CRP levels in blood will be measured.
Effect on indicators of Chronic inflammation (homocysteine) in blood | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on indicators of Indicators of Chronic inflammation in blood when compared to placebo and baseline. For this homocysteine levels in blood, will be measured.
Effect on indicators of Chronic inflammation (BDNF) in blood | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on indicators of Indicators of Chronic inflammation in blood when compared to placebo and baseline. For this BDNF (brain-derived neurotrophic factor protein) in blood will be measured.
Effect on indicators of Chronic inflammation (IL-11) in blood | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on indicators of Indicators of Chronic inflammation in blood when compared to placebo and baseline. For this IL-11 levels in blood will be measured.
Effect on indicators of Chronic inflammation (IL-6) in blood | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on indicators of Indicators of Chronic inflammation in blood when compared to placebo and baseline. For this, IL-6 levels in blood will be measured.
Effect on indicators of Chronic inflammation (IL-10) in blood | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on indicators of Indicators of Chronic inflammation in blood when compared to placebo and baseline. For this IL-10 levels in blood will be measured.
Effect on indicators of Chronic inflammation (TNF-α) in blood | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on indicators of Indicators of Chronic inflammation in blood when compared to placebo and baseline. For this TNF-α levels in blood will be measured.
Effect on indicators of Chronic inflammation in feces | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on indicators of Indicators of Chronic inflammation in feces when compared to placebo and baseline. For this Calprotectin levels in feces will be measured

OTHER OUTCOMES:
Effect on Musculoskeletal strength | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on the Musculoskeletal strength when compared to placebo and baseline. Musculoskeletal strength will measured by grip strength using a hand dynamometer (dominant arm) (expressed in kg).
Effect on Visual-motor coordination | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on Visual-motor coordination when compared to placebo and baseline. Visual-motor coordination of study participants (expressed in seconds) will be measured by the "Manipulation and Dexterity Test - Pegboard".
Effect on Indicators of general health and well-being | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on Indicators of general health and well-being when compared to placebo and baseline.
  The SF-12 will be used to assess general health and well-being: physical component summary and mental component summary scales (T score, expressed in a.u.). Lowest Value: 0, Highest Value: 100. A higher score means a better outcome,
Effect on Indicators of sleeping quality status | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on Indicators of sleeping quality status when compared to placebo and baseline.
  The PSQI global score will be used to assess sleep quality (expressed in a.u., range 0-21). Lowest Value: 0, Highest Value: 21. A higher score means a worse outcome
Effect on gastrointestinal function | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on gastrointestinal function when compared to placebo and baseline.
  The GSRS (Gastrointestinal Symptom Rating Scale) will be used to assess the participants' gastrointestinal function (5 subscores) (expressed in a.u., range 1-7)
Effect on Glycemic status (Blood insulin) | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on Glycemic status when compared to placebo and baseline. For this, blood Insulin levels will be measured.
Effect on Glycemic status (Glucose levels) | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on Glycemic status when compared to placebo and baseline. For this, blood glucose levels will be measured.
Effect on indicators of insulin resistance | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on insulin resistance when compared to placebo and baseline. For this (HOMA-IR technique) (expressed in a.u.) will be used.
Effect on Blood lipid levels | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on Blood lipid levels when compared to placebo (between group comparison) and baseline (within group comparison)
Effect on Body weight | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on Body weight when compared to placebo (between group comparison) and baseline (within group comparison)
Effect on Microbiome composition | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on Microbiome composition when compared to placebo and baseline. Microbiome composition will be measured using full shotgun sequencing.
Effect on Microbiome diversity | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on Microbiome diversity when compared to placebo and baseline. Microbiome diversity will be measured using full shotgun sequencing.
Effect on fecal metabolomic profile | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on fecal metabolomic profile when compared to placebo and baseline. Metabolomic profile will be analyzed using semi-polar liquid chromatography-mass spectrometry (LC-MS)/MS method.
Effect on Fecal organic acid levels | Timeframe - Day 0 (V2), Day 45 (V3) and Day 90 (V4)
  To assess the effect of 3 months of daily consumption of Humiome® Post LB on Fecal organic acid levels when compared to placebo (between group comparison) and baseline (within group comparison)

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Sadaghian, PhD, Study Director — DSM Nutritional Products, Inc.
Locations (1):
- analyze & realize GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No